CLINICAL TRIAL: NCT06484686
Title: An Open-label Clinical Trial to Evaluate the Immunity Persistence of Live Attenuated Varicella Vaccine At 6 and 10 Years After Booster Dose Immunization with Live Attenuated Varicella Vaccine
Brief Title: An Immunity Persistence Study of Booster Dose of Live Attenuated Varicella Vaccine
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac (Dalian) Vaccine Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO-VZV-4005
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Group (Experimental): Subjects will be collected venous blood at 6 and 10 years after booster immunization.
  Interventions: Biological: Live Attenuated Varicella Vaccine

INTERVENTIONS:
Biological: Live Attenuated Varicella Vaccine — lyophilized powder, subcutaneous injection

SUMMARY:
This an open-label phase Ⅳ clinical trial of live attenuated varicella vaccine manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd.The purpose of this study is to evaluate the immunity persistence of live attenuated varicella vaccine at 6 and 10 years after booster dose.

DETAILED DESCRIPTION:
A total of 792 subjects aged 2 to 6 years including in per-protocol set (PPS) of immunogenicity assessment from previous phase Ⅲ clinical trial were enrolled. About 3.0ml of venous blood was collected at 6 and 10 years after booster immunization for antibody detection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in PPS of previous phase Ⅲ clinical trial of varicella vaccine;
* The subjects and/or guardian can understand and voluntarily sign the informed consent form;
* Proven legal identity.

Exclusion Criteria:

* Beyond the blood collection window period;
* History of varicella or shingles;
* History of varicella vaccination since phase Ⅲ clinical trial;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 414 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Seropositive rate | at 6 years after booster vaccination
  The seropositive rate of varicella-zoster virus (VZV) antibodies at 6 years after booster vaccination
Seropositive rate | at 10 years after booster vaccination
  The seropositive rate of VZV antibodies at 10 years after booster vaccination
GMT of VZV antibody | at 6 years after booster vaccination
  The GMT of VZV antibodies at 6 years after booster vaccination
GMT of VZV antibody | at 10 years after booster vaccination
  The GMT of VZV antibodies at 10 years after booster vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Lili Huang, Principal Investigator — Henan Provincial Center for Disease Control and Prevention
Locations (1):
- Henan Provincial Center for Disease Control and Prevention, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No